CLINICAL TRIAL: NCT03498326
Title: Gemcitabine and Celecoxib Combination Therapy in Treating Patients With R0 Resection Pancreatic Cancer
Acronym: GCRP
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Liang Tingbo, Chairman of Department of Hepatobiliary & Pancreatic Surgery, Vice president of the Second Affiliated Hospital, Zhejiang University School of Medicine, Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAHZhejiangU-GCRP
Record Dates: First submitted 2018-04-02; First posted 2018-04-13 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Pancreatic Cancer; Chemotherapy Effect
Keywords: pancreatic cancer; gemcitabine; celecoxib; R0 resection
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- gemcitabine (Experimental): one group patients receive the standard gemcitabine treatment at 1,8,15 of the chemotherapy cycle after R0 resection.
  Interventions: Drug: Gemcitabine
- gemcitabine plus celecoxib (Experimental): the other group patients receive the standard gemcitabine treatment at 1,8,15 of the chemotherapy cycle after R0 resection, and receive additional celecoxib every days during chemotherapy period.
  Interventions: Drug: Gemcitabine

INTERVENTIONS:
Drug: Gemcitabine — One group patients receive the standard gemcitabine treatment at 1,8,15 of the chemotherapy cycle after R0 resection at 1000mg/m2.
  Arms: gemcitabine
Drug: Gemcitabine — the other group patients receive the standard gemcitabine treatment at 1,8,15 of the chemotherapy cycle after R0 resection at 1000mg/m2, and receive additional celecoxib 200mg bid every days during chemotherapy period.
  Other Names: celecoxib
  Arms: gemcitabine plus celecoxib

SUMMARY:
The prognosis of pancreatic cancer is extremely poor, even in those patients who had underwent surgery, the 5-year survival is still less than 10%. Current guidelines recommend Gemcitabine monotherapy for R0 resection of pancreatic cancer. Inflammation plays an critical role in the development and progression of pancreatic cancer. Here we intend to assess the synergistic effect of using celecoxib in combination with gemcitabine on the treatment of R0 resection of pancreatic cancer.

DETAILED DESCRIPTION:
We choose those patients who had underwent the R0 resection of pancreatic ductal adenocarcinoma patients, and divided them into two groups randomly, one group patients were given gemcitabine only according the current guidelines, while the other group patients were given gemcitabine combined with the anti-inflammation agent Celecoxib. The disease free survivals, drugs related side effects, overall survivals and other endpoints events were recorded and analyzed, to assess the celecoxib could or couldn't synergist the gemcitabine anti tumor effect on R0 resection pancreatic cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old and above.
2. Surgery for R0 resection.
3. The gemcitabine chemotherapy regimen was not previously used for the treatment of other malignancies.
4. Eastern Cooperative Oncology Group score 0-2 points.
5. Blood routine: The neutrophil count is at least 1.5*10^9/ml, and the platelet count is at least 100*10^9/ml.Hemoglobin is at least 80g/L.
6. Liver function: bilirubin does not exceed 1.5 times the upper limit of normal; alanine aminotransferase and aspartate aminotransferase does not exceed the upper limit of normal 3 times; kidney function: creatinine ≤ 1.2 mg/dL.

Exclusion Criteria:

1. Endocrine carcinoma, acinar pancreatic carcinoma, or cystadenocarcinoma (cystadenocarcinoma).
2. Surgery for pancreatic cancer fails to reach the R0 resection criteria.
3. Pancreatic cancer received radiotherapy before surgery.
4. Malignant brain metastases.
5. There are other serious cancer history.
6. Active infection, severe diarrhea.
7. Others: Those who are allergic to celecoxib; or who are intolerant to celecoxib, require continuous aspirin or Non-steroidal anti-inflammatory drugs; similar chemical or biological components and sulfa drugs that constitute the study drug History of allergies; allergies, asthma, and rubella after taking aspirin or non-steroidal anti-inflammatory drugs; pregnancy or breastfeeding; active gastrointestinal ulcer/hemorrhage/perforation; Severe mental illness; severe heart failure; past serious cardiovascular thrombotic adverse events, severe hypertensive patients.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2018-04-02 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
disease free survival | Up to approximately 60 months
  the duration between the date of surgery and the date of disease relapse

SECONDARY OUTCOMES:
overall survival | Up to approximately 60 months
  the duration between the date of surgery and the date of patient death
Carbohydrate antigen 19-9 | Up to approximately 36 months
  serum Carbohydrate antigen 19-9 level
Quality of Life | Up to approximately 60 months
  assessed by the European Organization for Research and Treatment of Cancer Quality of Life-pancreatic cancer 26 score
Common Toxicity Criteria for Adverse Effects | Up to approximately 12 months
  according to Common Toxicity Criteria for Adverse Effects version 4

CONTACTS AND LOCATIONS:
Locations (1):
- the second affiliated hospital of Zhejiang University, Hangzhou, Zhejiang, China